CLINICAL TRIAL: NCT03878693
Title: The Effect of 4-methylpyrazole on Oxidative Metabolism of Acetaminophen in Healthy Volunteers
Brief Title: 4-methylpyrazole and Acetaminophen Metabolism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1805526976
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2018-06

CONDITIONS: Healthy Adult Volunteers
MeSH Terms: interventions — Fomepizole; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): Oral APAP and IV Fomepizole.
  Interventions: Drug: Fomepizole; Drug: APAP
- B (Active Comparator): Oral APAP.
  Interventions: Drug: APAP

INTERVENTIONS:
Drug: Fomepizole — IV 4-MP.
  Arms: A
Drug: APAP — Oral APAP

SUMMARY:
Oxidative metabolism of APAP will be studied with and without 4-MP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No APAP use in previous 2 weeks
* No ingestion of alcohol or drugs that affect CYP 2E1 over previous 5 days
* No allergy to APAP or fomepizole
* BMI < 29

Exclusion Criteria:

* Pregnant or lactating
* History of alcohol abuse
* Allergy to APAP or fomepizole
* Screening LFTs above normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Oxidative metabolism of APAP | 24 hours
  Measurement of oxidized metabolites of APAP

CONTACTS AND LOCATIONS:
Locations (1):
- BUMCP - Department of Medical Toxicology, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Kang AM, Padilla-Jones A, Fisher ES, Akakpo JY, Jaeschke H, Rumack BH, Gerkin RD, Curry SC. The Effect of 4-Methylpyrazole on Oxidative Metabolism of Acetaminophen in Human Volunteers. J Med Toxicol. 2020 Apr;16(2):169-176. doi: 10.1007/s13181-019-00740-z. Epub 2019 Nov 25. PMID 31768936